CLINICAL TRIAL: NCT02025790
Title: A Prospective Trial Comparing POEM to Pneumatic Dilatation for Treatment of Achalasia Cardia
Brief Title: POEM Versus Pneumatic Dilatation in Achalasia Cardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Nageshwar Reddy D, Chairman, Asian Institute of Gastroenterology, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG-POEM-01
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Achalasia Cardia
Keywords: Achalasia; POEM; Pneumatic dilatation; Eckardt score
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - POEM (Experimental): Per Oral Endoscopic Myotomy for treatment of achalasia
  Interventions: Procedure: Per Oral Endoscopic Myotomy (POEM)
- Group B - Dilatation (Active Comparator): - Pneumatic dilatation using a balloon for treatment of achalasia.
  Interventions: Procedure: Pneumatic Dilatation

INTERVENTIONS:
Procedure: Per Oral Endoscopic Myotomy (POEM) — * Mucosal incision - After submucosal injection, a 2-cm longitudinal mucosal incision is made at approximately 12 cm proximal to the gastroesophageal junction (GEJ).
  * Submucosal tunneling. A long submucosal tunnel is created to 3 cm distal to the GEJ.
  * Endoscopic myotomy is begun at 3 cm distal to the mucosal entry point, and is carried out in a proximal to distal direction to a total length of 10 cm.
  * Long endoscopic myotomy is performed 10 cm proximal to GEJ extending
  * Closure of mucosal entry: the mucosal incision is closed using hemostatic clips
  Arms: Group A - POEM
Procedure: Pneumatic Dilatation — Pneumatic dilatation using a Rigiflex balloon up to 35 mm at 8 psi for 1 minute.
  Arms: Group B - Dilatation

SUMMARY:
The aim of this study is to compare efficacy of POEM and pneumatic dilatation in treatment of achalasia cardia.

DETAILED DESCRIPTION:
Achalasia is an esophageal motility disorder which involves smooth muscle of the esophagus and the lower esophageal sphincter (LES). Achalasia causes difficulty swallowing, regurgitation, and sometimes chest pain and weight loss. Endoscopic treatments of achalasia can be provided in the form of dilatation of the LES or cutting of muscle fibers (myotomy) of the esophagus and of the LES under endoscopic viewing. Dilatation in this trial is accomplished with rigiflex balloons and myotomy via Per Oral Endoscopic Myotomy (POEM). The effectiveness of treatment of achalasia using each method will be compared in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Achalasia with Eckardt score at least 3 (0-12 scale achalasia least-most severe)
2. Age 18-75 years
3. Willing and able to comply with the study procedures and provide written informed consent form to participate in the study written informed consent form to participate in the study

Exclusion Criteria:

1. Severe comorbid illness
2. Previous esophageal or gastric surgery
3. Pseudo achalasia
4. Achalasia with esophageal diverticula
5. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 3 months post procedure
  Clinical success defined as reduction of Eckardt score (0-12 scale achalasia least-most severe) of achalasia to an Eckardt score of 3 or less post procedure

SECONDARY OUTCOMES:
Adverse events | 1 week post procedure
  All dilatation or POEM related adverse events, including type, required intervention, severity, time to resolution

OTHER OUTCOMES:
Cytokine levels | Pre procedure and immediately and 6 hours post procedure
  Post procedural inflammation compared to baseline as measured by blood cytokine levels
Long term clinical success | 6 and 12 months post procedure
  Long term clinical success at 6 and 12 months post procedure compared to baseline.
LES pressure | 3, 6 and12 months post procedure
  Post procedure reduction in LES pressure at 3, 6 and 12 months compared to baseline.
Quality of life | 3, 6 and 12 months post procedure
  Quality of Life (QOL) improvement at 3, 6 and 12 months post procedure compared to baseline using SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: D Nageshwar Reddy, MD, Principal Investigator — Asian Institute of Gastroenterology (AIG)
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India